CLINICAL TRIAL: NCT00717197
Title: Pilot Study to Determine Therapeutic Response of Oral Capecitabine (Xeloda) in Recurrent High Grade Gliomas (HGGs) by Establishing the Radiographic Response Rate Using Modified Macdonald Criteria
Brief Title: Study of Capecitabine to Treat Recurrent High Grade Gliomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HGG-001
Record Dates: First submitted 2008-07-15; First posted 2008-07-17 (Estimated); Results first posted 2013-03-25 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-06

CONDITIONS: Malignant Glioma
Keywords: HGG; anaplastic astrocytoma; anaplastic oligodendroglioma; anaplastic mixed glioma; glioblastoma multiforme; GBM; Xeloda; capecitabine
MeSH Terms: conditions — Glioma; Astrocytoma; Oligodendroglioma; Glioblastoma | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Capecitabine (Experimental): Capecitabine (1,000-1,250 mg/m2) taken by mouth twice daily for 14 out of 21 consecutive days until progression or unacceptable toxicity.
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Capecitabine — 1,000-1,250 mg/m2 taken by mouth twice daily for 14 out of 21 consecutive days until progression or unacceptable toxicity.
  Other Names: Xeloda

SUMMARY:
The purpose of this study is to determine if capecitabine is effective in the treatment of high grade gliomas that have returned after completing treatment.

DETAILED DESCRIPTION:
High grade gliomas (HGGs) represent a heterogenous group of primary brain tumors that share WHO grade III or IV classification (anaplastic astrocytoma, anaplastic oligodendroglioma, anaplastic mixed glioma, and glioblastoma multiforme). Despite the upfront use of surgery, radiation, and chemotherapy, high grade gliomas uniformly result in recurrence and death. Palliative chemotherapy offers an improvement in time to progression, symptom control, quality of life, and potential survival; however, no established chemotherapy regimen for recurrence exists and new treatments are needed. Oral capecitabine is a rationale strategy for therapeutic palliation of recurrent high grade gliomas given its oral administration, its well-known kinetics and toxicities, its non-competitive toxicities to other high grade glioma treatments, its well established management algorithms, its established evidence of entry into the central nervous system, and its evidence of safety and efficacy in malignancies in the central nervous system.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of high grade glioma (WHO grade III or IV: anaplastic astrocytoma, anaplastic oligodendroglioma, anaplastic mixed glioma, and glioblastoma multiforme)
* Male or female 18 years of age or older
* Negative pregnancy test (if of childbearing potential)
* Any number of previous recurrences will be allowed
* Karnofsky Performance Status > 60
* Hematocrit > 30,000
* White blood cell count > 1,500
* Platelet > 100,000
* Absolute Neutrophil Count > 1,000
* Bilirubin < 1.5 x upper limits of normal
* Transaminases (ALT and AST) < 1.5 x upper limits of normal
* Creatinine < 1.5 x upper limits of normal
* Adequate medical health to participate in this study
* Adequate documentation of menopause (natural/surgical) or patient commitment to routine use of reliable birth control (barrier/hormonal)
* Ability to read and understand the informed consent document
* Ability and willingness to follow all requirements of the study including following all directions, taking medication as prescribed and completing all diaries and forms

Exclusion Criteria:

* Karnofsky Performance Status < 60
* Hematocrit < 30,000
* White blood cell count < 1,500
* Platelet < 100,000
* Absolute Neutrophil Count < 1,000
* Bilirubin >1.5 x upper limits of normal
* Transaminases (ALT and AST) > 1.5 x upper limits of normal
* Creatinine > 1.5 x upper limits of normal
* Inability to undergo gadolinium-contrasted MRIs, including severe claustrophobia or insufficient allergy prophylaxis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-07; Primary Completion 2012-03 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin Dunbar, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the investigator's clinical practice from October 2008 thru June 2011.
Pre-assignment Details: 30 participants were enrolled in the study. 7 were excluded from participation prior to group assignment [5 were unable to purchase study drug; 1 had rapid tumor growth; and, 1 was withdrawn by the investigator for mental health reasons].
Groups:
- Capecitabine: Capecitabine (1,000-1,250 mg/m2) was taken by mouth twice daily for 14 out of 21 consecutive days until disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Capecitabine
Started | 30
Completed | 23
Not Completed | 7
Not completed — Unable to purchase study drug | 5
Not completed — Tumor Progression | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Capecitabine
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 7
Age Continuous [Mean (Standard Deviation); unit: years] | 51.5 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Progression-free Survival.
Description: Gadolinium-contrasted MRIs were used to assess radiographic response every 2 cycles (~6 weeks). Tumor progression was defined by increasing tumor size, new areas of tumor, or unequivocal neurologic deterioration.
Time Frame: From date of first dose of study drug until month 6.
Population: Per protocol
Measure: Number (95% Confidence Interval); unit: percentage of participants with PFS6
Arm/Group | Capecitabine
Number analyzed (Participants) | 23
percentage of participants with PFS6 | 21.7 [7.46 to 43.7]
Statistical Analysis 1: Comparison: Capecitabine; Test type: Superiority or Other; Percentage = 21.7, 95% CI 2-sided [7.46 to 43.7], Standard Error of Mean 7.27

ADVERSE EVENTS:
Time Frame: Adverse events were collected beginning with the first dose of study drug and continuing until 14 days after the last dose of study drug.
Arm/Group | Capecitabine
Serious Adverse Events (participants affected / at risk) | 21/23
Other Adverse Events (participants affected / at risk) | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Capecitabine (N=23)
Mental Status (Nervous system disorders) | 4
Death (General disorders) | 21 (21)
Fever (General disorders) | 1
Gait (Musculoskeletal and connective tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Dairrhea (Gastrointestinal disorders) | 1
Ataxia (Nervous system disorders) | 1
Levetiracetam, Low Level (General disorders) | 1
Phenytoin, High Level (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Capecitabine (N=23)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
ALT (Metabolism and nutrition disorders) | 4
Mood Alteration (Nervous system disorders) | 4
Speech Impairement (Nervous system disorders) | 2
AST (Metabolism and nutrition disorders) | 3
Ataxia (Nervous system disorders) | 2
Bilirubin (Metabolism and nutrition disorders) | 1
Blindness (Eye disorders) | 1
Blurred Vision (Eye disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Cholesterol (Metabolism and nutrition disorders) | 1
Cognitive Disturbance (Nervous system disorders) | 1
Confusion (Nervous system disorders) | 2
Constipation (Gastrointestinal disorders) | 6
Diarrhea (Gastrointestinal disorders) | 6
Dizziness (Nervous system disorders) | 1
Dysphagia (Gastrointestinal disorders) | 3
Edema (General disorders) | 4
Fatigue (General disorders) | 10
Hyperglycemia (Metabolism and nutrition disorders) | 5
Hand-foot Skin Reaction (Skin and subcutaneous tissue disorders) | 5
Heartburn (Gastrointestinal disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 4
Headache (Nervous system disorders) | 4
Infection (Infections and infestations) | 3
Insomnia (General disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 3
Lymphopenia (Blood and lymphatic system disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 4
Neuropathy (Nervous system disorders) | 8
Pain (General disorders) | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Platelets (Blood and lymphatic system disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Seizure (Nervous system disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 2
Leukocytes (Blood and lymphatic system disorders) | 2
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1
Somnolence (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes